CLINICAL TRIAL: NCT05327244
Title: The Impact of Real-World Vibration Feedback Gait Retraining on Gait Biomechanics in People With Chronic Ankle Instability
Acronym: RWVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Academy of Orthopaedic Physical Therapy (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-0399
Record Dates: First submitted 2022-04-06; First posted 2022-04-14 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Chronic Ankle Instability
Keywords: ankle; walking; biofeedback

STUDY DESIGN:
Intervention Model Description: All CAI participants will be assigned to the intervention arm and will all receive the same treatment (6 sessions of RWVF gait retraining in 2-weeks). Posttest data from CAI participants in arm 1 will be compared to data from pre-collected de-identified healthy control data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): All CAI participants will complete the same intervention and will walk 6, 1-mile paths in the real wold (ie: around campus) with vibration feedback within 2 weeks of baseline assessment. A study team member will accompany each participant during each training.
  Interventions: Other: Real-world vibration feedback gait retraining
- Healthy Control (No Intervention): Posttest data from CAI participants will be compared to de-identified healthy control data collected as part of a previous study. Healthy control participants completed a single research session to collect walking biomechanics using the same methods as this project. They received no further follow up or intervention and the inclusion/ exclusion criteria for this group match those of the chronic ankle instability cohort.

INTERVENTIONS:
Other: Real-world vibration feedback gait retraining — Participants will walk with a vibration feedback tool attached to their shoelaces. A small force sensing resistor is taped to the foot bed of the shoe under the lateral foot and a vibration motor is placed over the outside of the ankle with a strap. When a participant walks on the outside of their foot, they will exceed the pressure threshold and activate the feedback which signifies an incorrect foot placement. The feedback is intended to prompt a correct foot placement on the subsequent step. Participants will use the same feedback tool for 6 real world training sessions.
  Arms: Intervention

SUMMARY:
People with chronic ankle instability (CAI) demonstrate altered gait or walking mechanics which cause people to walk on the outside of their foot and increases the risk of additional ankle sprains, abnormal cartilage strain, and early joint degeneration. Evidence indicates that common treatments for CAI do not impact gait, leaving unresolved impairments that can lead to lifelong disability. Recent lab-based gait retraining with visual and auditory feedback has immediately improved walking mechanics. However, real-world training is hypothesized to generate long-term changes by incorporating short, frequent training sessions over a variety of surfaces. These are key training parameters to produce lasting change. Pilot data using real-world vibration feedback (RW-VF) suggest that a single session immediately improves walking mechanics with changes lasting for up to 5 minutes. Despite promising initial results, there remains a critical need to determine the impact of multiple RW-VF sessions as an initial step to developing a protocol capable of long-term improvements. The purpose of this proposal is to determine the extent to which 2-weeks of RW-VF restores gait biomechanics in those with CAI. Twenty people with CAI will be enrolled and complete a two-week gait retraining protocol with vibration feedback. Walking mechanics before, immediately after, and 1 week and 4 weeks following the training will be compared. These contributions can be significant as positive results will support a paradigm shift in treatments for people with CAI and lay the foundation for large scale clinical trials aimed at optimizing long term gains. The outcomes of future research have the potential to advance evidenced based rehabilitation interventions not only for people with CAI but also for people who have sustained a variety of musculoskeletal injuries as there is strong evidence that other lower extremity pathologies cause lifelong limitations, including changes in walking mechanics which lead to degenerative changes to other joints.

DETAILED DESCRIPTION:
Background: There are 3.1 million lateral ankle sprains in the United States per year, of which about 40% will develop persistent limitations leading to chronic ankle instability (CAI). People with CAI demonstrate altered walking gait mechanics including increased inversion (ie: the foot rolling outward) and a lateral shift in the location of the center of pressure (COP) under the foot. These changes cause people to walk on the outside of their foot and increases the risk for additional ankle sprains, abnormal cartilage strain, and early post traumatic ankle arthritis (PTOA). Evidence indicates that common treatments for CAI do not impact gait, leaving unresolved impairments that can lead to lifelong disability. Recently walking with novel sensory feedback techniques (visual, auditory, and visual stimuli) has immediately improved walking mechanics during laboratory training. However, real-world (RW) training is hypothesized to generate long-term changes by incorporating short, frequent training sessions over a variety of surfaces which are key training parameters to produce lasting change. Vibration feedback (VF) is currently the only tool capable of being deployed in the real world. Recent pilot data suggest that a single VF training session in the RW immediately improves ankle and COP position with changes lasting for up to 5 minutes. Despite these promising initial results, there remains a critical need to determine the impact of multiple real-word vibration feedback (RW-VF) sessions as an initial step to developing a protocol capable of long-term improvements.

Purpose: The purpose of this proposal is to examine the effectiveness of a new treatment approach by determining the extent to which 2-weeks of RW-VF restores gait biomechanics in those with CAI.

Design: Cohort Study Methods: Kinematic and kinetic data will be captured from 20 participants with CAI at two baseline training sessions within 48 hours of each other (B1 and B2) while the participant walks on an instrumented treadmill. These data will be used to calculate the minimal detectable change (MDC), which is the stability of the walking measures. Following B2, participants will be fitted with the VF tool and complete the first of six training sessions. During training sessions, participants will walk six standardized but unique 1-mile RW routes with VF within a two-week time period. The order of the routes will be determined by a random number generator. Three additional biomechanical walking assessments will be completed within 72 hours of (P-2), one week following the final training (F-1), and 4 weeks following the final training (F-4).

Data Analysis: The primary analysis will determine the impact of RW-VF on COP location during the stance phase of walking in people with CAI. COP location will be compared before and after treatment (B1:P-2) using paired t-tests to determine the immediate impact of RW-VF training. The change between B1 and P-2 will be compared to the MDC to rule out measurement error. Next, COP location between B1 and F-1, and B1 and F-4 will be calculated to determine the extent to which the COP change is retained and compared to the MDC to rule out measurement error. Finally, COP data from posttest and retention timepoints will be compared to a database of walking biomechanics data from healthy controls using independent t-tests to determine similarities between people with and without CAI following training. The secondary analysis will repeat the primary using ankle position in the frontal plane (inversion/ eversion) during stance.

Significance: These contributions have the potential to be significant because positive results will support a paradigm shift in treatments for people with CAI. Positive results will also lay the foundation for large scale clinical trials comparing the current standard of care to the standard of care with the addition of RW-VF training to optimize long term gains. The outcomes of future research have the potential to advance evidenced based rehabilitation interventions not only for people with CAI but also for people who have sustained a variety of musculoskeletal injuries as there is strong evidence that other lower extremity pathologies cause lifelong limitations, including changes in walking mechanics which lead to degenerative changes to other joints.

ELIGIBILITY:
CAI group:

Inclusion Criteria:

* between the ages of 18 - 35 years
* will have a history of at least 1 significant lateral ankle sprain which occurred at least 12 months prior to enrollment defines as a sprain which caused at least 1 day of interrupted physical activity
* have a history of recurrent sprains and/or episodes of "giving way"
* have a sense of ankle instability measured by a score of ≥ 11 on the Identification of Functional Ankle Instability (IdFAI)
* have self-reported functional limitations measured by a score of < 90% of the Foot and Ankle Ability Measure (FAAM)-Activities of Daily Living subscale and < 80% on the FAAM-Sport subscale.

Exclusion Criteria:

* evidence of bilateral CAI using the criteria above
* history of previous surgery in either lower extremity
* history of a fracture requiring realignment in either lower extremity
* an acute (< 12 weeks from enrollment) injury to either lower extremity
* any condition known to affect gait such as peripheral neuropathy, diabetes, neurological disorders, or neurodegenerative diseases
* knowingly pregnant.

Criteria for precollected healthy control data Inclusion/ Exclusion Criteria

* between the ages of 18-35 years
* no previous history of lower extremity surgery
* no lower extremity injury history in the past 6 months
* no history of neurological disorders (i.e.: stroke, cerebral palsy, multiple sclerosis, etc.)
* not knowingly pregnant. Patient reported outcomes (ie: FAAM, IdFAI) were not collected as part of the previous study, therefore cannot be used as inclusion or exclusion criteria.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Immediate and retained changes in the center of pressure location under the foot at initial contact within the chronic ankle instability group in response to 2-weeks of RWVF gait retraining. | COP location during walking will be measured at baseline, within 72 hours of completing the intervention (P-2), 1 week after the intervention (F-1), 1 month after the intervention (F-4).
  The location of the center of pressure (COP) under the foot will be collected while participants walk for 1-minute on an instrumented treadmill at each assessment in this repeated measures study (baseline, P-2, F-1, F-4). Data from each stance phase of walking will be divided into 10 equal parts each representing 10% of stance and averaged across all steps. Subphase 1 of the data will be used for the primary outcome as it represents initial contact of gait.

SECONDARY OUTCOMES:
Immediate and retained changes in the center of pressure location under the foot from 20% to 100% of the walking stance phase within the chronic ankle instability group in response to 2-weeks of RWVF gait retraining. | COP location during walking will be measured at baseline, within 72 hours of completing the intervention (P-2), 1 week after the intervention (F-1), 1 month after the intervention (F-4).
  The location of the COP under the foot will be collected while participants walk for 1-minute on an instrumented treadmill at each assessment in this repeated measures study (baseline, P-2, F-1, F-4). Data from each stance phase of walking will be divided into 10 equal parts each representing 10% of stance and averaged across all steps. Subphases 2-10 of the data will be used for this secondary outcome.
Differences between the COP location in people with CAI following 2-weeks of RWVF gait retraining and the COP location in healthy controls. | The COP location during walking will be measured following 2-weeks of training (P-2) in the CAI cohort and compared to pre-collected, de-identified healthy control data from a single session.
  The location of the COP under the foot will be collected while CAI participants walk for 1-minute on an instrumented treadmill following 2-weeks of RWVF gait retraining (P-2). Previously, data were collected during 1-minute of walking on an instrumented treadmill from a healthy control cohort. Data from each stance phase of walking from both groups will be divided into 10 equal parts each representing 10% of stance and averaged across all steps. Subphases 1-10 of the data will be used for this secondary outcome to compare the COP location between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Kimmery Migel, PT, DPT, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: starting 9 months and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Waterman BR, Owens BD, Davey S, Zacchilli MA, Belmont PJ Jr. The epidemiology of ankle sprains in the United States. J Bone Joint Surg Am. 2010 Oct 6;92(13):2279-84. doi: 10.2106/JBJS.I.01537. PMID 20926721
- [Background] Gribble PA, Delahunt E, Bleakley CM, Caulfield B, Docherty CL, Fong DT, Fourchet F, Hertel J, Hiller CE, Kaminski TW, McKeon PO, Refshauge KM, van der Wees P, Vicenzino W, Wikstrom EA. Selection criteria for patients with chronic ankle instability in controlled research: a position statement of the International Ankle Consortium. J Athl Train. 2014 Jan-Feb;49(1):121-7. doi: 10.4085/1062-6050-49.1.14. Epub 2013 Dec 30. PMID 24377963
- [Background] Wikstrom EA, Song K, Tennant JN, Dederer KM, Paranjape C, Pietrosimone B. T1rho MRI of the talar articular cartilage is increased in those with chronic ankle instability. Osteoarthritis Cartilage. 2019 Apr;27(4):646-649. doi: 10.1016/j.joca.2018.12.019. Epub 2019 Jan 8. PMID 30634032
- [Background] Gribble PA, Bleakley CM, Caulfield BM, Docherty CL, Fourchet F, Fong DT, Hertel J, Hiller CE, Kaminski TW, McKeon PO, Refshauge KM, Verhagen EA, Vicenzino BT, Wikstrom EA, Delahunt E. Evidence review for the 2016 International Ankle Consortium consensus statement on the prevalence, impact and long-term consequences of lateral ankle sprains. Br J Sports Med. 2016 Dec;50(24):1496-1505. doi: 10.1136/bjsports-2016-096189. Epub 2016 Jun 3. PMID 27259753
- [Background] Torp DM, Thomas AC, Donovan L. External feedback during walking improves measures of plantar pressure in individuals with chronic ankle instability. Gait Posture. 2019 Jan;67:236-241. doi: 10.1016/j.gaitpost.2018.10.023. Epub 2018 Oct 21. PMID 30380508
- [Background] Donovan L, Feger MA, Hart JM, Saliba S, Park J, Hertel J. Effects of an auditory biofeedback device on plantar pressure in patients with chronic ankle instability. Gait Posture. 2016 Feb;44:29-36. doi: 10.1016/j.gaitpost.2015.10.013. Epub 2015 Oct 27. PMID 27004629
- [Background] Feger MA, Hertel J. Surface electromyography and plantar pressure changes with novel gait training device in participants with chronic ankle instability. Clin Biomech (Bristol). 2016 Aug;37:117-124. doi: 10.1016/j.clinbiomech.2016.07.002. Epub 2016 Jul 7. PMID 27423026
- [Background] Yen SC, Corkery MB, Donohoe A, Grogan M, Wu YN. Feedback and Feedforward Control During Walking in Individuals With Chronic Ankle Instability. J Orthop Sports Phys Ther. 2016 Sep;46(9):775-83. doi: 10.2519/jospt.2016.6403. Epub 2016 Aug 5. PMID 27494057
- [Background] Feger MA, Hart JM, Saliba S, Abel MF, Hertel J. Gait training for chronic ankle instability improves neuromechanics during walking. J Orthop Res. 2018 Jan;36(1):515-524. doi: 10.1002/jor.23639. Epub 2017 Aug 11. PMID 28653780
- [Background] Erhart-Hledik JC, Asay JL, Clancy C, Chu CR, Andriacchi TP. Effects of active feedback gait retraining to produce a medial weight transfer at the foot in subjects with symptomatic medial knee osteoarthritis. J Orthop Res. 2017 Oct;35(10):2251-2259. doi: 10.1002/jor.23527. Epub 2017 Feb 9. PMID 28120496
- [Background] Migel KG, Wikstrom EA. The effect of laboratory and real world gait training with vibration feedback on center of pressure during gait in people with chronic ankle instability. Gait Posture. 2021 Mar;85:238-243. doi: 10.1016/j.gaitpost.2021.02.011. Epub 2021 Feb 17. PMID 33621942
- [Background] Migel KG, Wikstrom EA. Immediate effects of vibration biofeedback on ankle kinematics in people with chronic ankle instability. Clin Biomech (Bristol). 2021 Dec;90:105495. doi: 10.1016/j.clinbiomech.2021.105495. Epub 2021 Sep 25. PMID 34601325